CLINICAL TRIAL: NCT03717259
Title: Recovery of Short-term Renal Function in Post-transplant Patients Living Donor: Comparison Between Graft Procurement Techniques - Open Surgery, Laparoscopic Assisted Hand and Pure Laparoscopic
Brief Title: Recovery of Short-term Renal Function in Post-transplant Patients Living Donor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Alejandro Gonzalez-Ojeda, Full time surgical researcher, Instituto Mexicano del Seguro Social
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Post_transplant_2016
Record Dates: First submitted 2018-06-26; First posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Nephrectomy
Keywords: Renal Donation; Renal Transplant; Open Nephrectomy; Laparoscopic Nephrectomy; Hand Assisted; Surgical Morbidity

STUDY DESIGN:
Intervention Model Description: This is an analytical cross-sectional study for which patients with terminal chronic kidney disease will be taken from kidney transplanted from a related live donor in a tertiary hospital. The selection of patients will be done with a non-probabilistic sampling of consecutive cases.
  Kidney transplantation from a live donor will be carried out by means of kidney graft procurement techniques using open surgery, laparoscopic hand-assisted surgery or pure laparoscopic surgery.
  The statistical analysis will be performed with Student´s t-test and Chi-square test. To determine if the intervening variables affected the postoperative renal function, we will perform a multivariate analysis. We will consider a significant P value when it is <0.05.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open nephrectomy (Active Comparator): These patients will undergo an open nephrectomy.
  Interventions: Procedure: Open nephrectomy
- Hand-assisted laparoscopic nephrectomy (Active Comparator): These patients will undergo a hand-assisted nephrectomy.
  Interventions: Procedure: Hand-assisted laparoscopic nephrectomy
- Laparoscopic nephrectomy (Active Comparator): These patients will undergo a pure laparoscopic nephrectomy.
  Interventions: Procedure: Laparoscopic nephrectomy

INTERVENTIONS:
Procedure: Open nephrectomy — The surgical technique for open nephrectomy consists of placing the donor in the lateral decubitus position and making an incision with or without rib resection that allows retroperitoneal access.
  Arms: Open nephrectomy
Procedure: Hand-assisted laparoscopic nephrectomy — The hand-assisted technique begins with the incision for the introduction port of the hand, the renal artery and vein are divided using endoscopic staples and the graft is manually removed.
  Arms: Hand-assisted laparoscopic nephrectomy
Procedure: Laparoscopic nephrectomy — In the pure laparoscopic technique the patient is placed in the same position of lateral decubitus and after introducing the trocars in the abdomen, the colon is mobilized and the renal capsule is divided, the kidney is removed after performing the cut of the renal artery and vein through a suprapubic incision.
  Arms: Laparoscopic nephrectomy

SUMMARY:
Objectives: To describe and analyze the perioperative and functional evolution of short-term renal graft in patients with kidney transplantation from a live donor, comparing three surgical techniques for obtaining kidney graft: open nephrectomy, laparoscopic hand-assisted nephrectomy, and pure laparoscopic nephrectomy.

DETAILED DESCRIPTION:
Analytical cross-sectional study that will compare the three renal graft procurement techniques: open nephrectomy, laparoscopic hand-assisted nephrectomy, and pure laparoscopic nephrectomy. The investigators will analyze serum creatinine values on days 1, 5 and 28 post renal transplantation. The operative, medical and surgical morbidity will also be evaluated, considering the bleeding in the donor, times of ischemia and the need for JJ catheter placement in the recipient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with terminal chronic kidney disease who will receive a kidney transplant in the transplant service of the National Medical Center of the West of living donor related to the means of obtaining the kidney graft by laparoscopic hand assisted or pure laparoscopic surgery.

Exclusion Criteria:

* Patients who for some reason can not find your complete medical record.
* Patients obtained a kidney graft from a brain death donor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of medical complications in renal graft recipients through 30 day after the nephrectomy. | Through 30 days post surgery.
  The investigators will evaluate the presence of surgical and medical complications in renal graft recipients obtained by open nephrectomy, hand assisted nephrectomy, and pure laparoscopic nephrectomy.

SECONDARY OUTCOMES:
Days of hospital stay | 30 days after the nephrectomy.
  Differences in the days of hospital stay of the renal donor comparing the techniques used to obtain the graft.
Bleeding during the nephrectomy | Through the nephrectomy
  The investigators will measure the volume of bleeding.
JJ catheter placement | Perioperative (5 days post surgery)
  The investigators will describe the number of patients who underwent a JJ catheter.
Serum creatinine | Days post trasplant 1, 5 and 28.
  Measurement of serum creatinine in kidney transplant patients.
Duration of the nephrectomy in minutes | Minutes from the beginning to the end of the nephrectomy
  The investigators will measure how long the nephrectomies lasts
Warm ischemia time in the graft | Time in minutes between the clamping of the renal vessels and the cooling of the graft with the preservation liquid at 4º C
  The investigators will measure the time of warm ischemia during nephrectomy

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Sánchez Martínez, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Roberto Martínez De Pinillos Valverde, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Eduardo González-Espinoza, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Clotilde Fuentes Orozco, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Roberto Mares País, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Francisco José Barbosa Camacho, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Diego Andrés Gallardo Vega, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Alejandro González Ojeda, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villeda-Sandoval CI, Rodriguez-Covarrubias F, Cortes-Aguilar G, Alberu-Gomez J, Vilatoba-Chapa M, Sotomayor M, Feria-Bernal G, Gabilondo F, Gabilondo-Pliego B. Hand-assisted laparoscopic versus open donor nephrectomy: a retrospective comparison of perioperative and functional results in a tertiary care center in Mexico. Transplant Proc. 2013 Nov;45(9):3220-4. doi: 10.1016/j.transproceed.2013.03.055. PMID 24182788
- [Background] Altinel M, Akinci S, Gunes ZE, Olcucuoglu E, Gonenc F, Yazicioglu AH. Open versus laparoscopic donor nephrectomy: perioperative parameters and graft functions. Transplant Proc. 2011 Apr;43(3):781-6. doi: 10.1016/j.transproceed.2011.01.113. PMID 21486597
- [Background] Chin EH, Hazzan D, Edye M, Wisnivesky JP, Herron DM, Ames SA, Palese M, Pomp A, Gagner M, Bromberg JS. The first decade of a laparoscopic donor nephrectomy program: effect of surgeon and institution experience with 512 cases from 1996 to 2006. J Am Coll Surg. 2009 Jul;209(1):106-13. doi: 10.1016/j.jamcollsurg.2009.02.060. Epub 2009 May 1. PMID 19651070
- [Background] Rojas-Manjarrez MA, Fernandez-Diaz OF, Sandoval-Sandoval MJ, Valdespino-Mejia C, Monteon-Ramos F, Gonzalez-Ojeda A. [Urological complications after kidney transplantation]. Cir Cir. 2008 Mar-Apr;76(2):133-7. Spanish. PMID 18492434
- [Background] Perez Fentes DA, Blanco Parra M, Toucedo Caamano V, Romero Burgos R, Punal Rodriguez JA, Varo Perez E. [Surgical complications after kidney transplantation. Research based on 185 cases]. Actas Urol Esp. 2005 Jun;29(6):578-86. doi: 10.1016/s0210-4806(05)73300-3. Spanish. PMID 16092682
- [Background] Wolf JS Jr, Tchetgen MB, Merion RM. Hand-assisted laparoscopic live donor nephrectomy. Urology. 1998 Nov;52(5):885-7. doi: 10.1016/s0090-4295(98)00389-6. PMID 9801121
- [Background] Kalble T, Lucan M, Nicita G, Sells R, Burgos Revilla FJ, Wiesel M; European Association of Urology. EAU guidelines on renal transplantation. Eur Urol. 2005 Feb;47(2):156-66. doi: 10.1016/j.eururo.2004.02.009. PMID 15661409
- [Background] Emery DL, Rothel JS, Wood PR. Influence of antigens and adjuvants on the production of gamma-interferon and antibody by ovine lymphocytes. Immunol Cell Biol. 1990 Apr;68 ( Pt 2):127-36. doi: 10.1038/icb.1990.18. PMID 2116995
- [Background] Stifelman MD, Hull D, Sosa RE, Su LM, Hyman M, Stubenbord W, Shichman S. Hand assisted laparoscopic donor nephrectomy: a comparison with the open approach. J Urol. 2001 Aug;166(2):444-8. doi: 10.1016/s0022-5347(05)65960-5. PMID 11458044
- [Background] Nogueira JM, Cangro CB, Fink JC, Schweitzer E, Wiland A, Klassen DK, Gardner J, Flowers J, Jacobs S, Cho E, Philosophe B, Bartlett ST, Weir MR. A comparison of recipient renal outcomes with laparoscopic versus open live donor nephrectomy. Transplantation. 1999 Mar 15;67(5):722-8. doi: 10.1097/00007890-199903150-00014. PMID 10096529
- [Background] Meyer F, Nichele SA, Adamy A, Santos LS, Machado C. Early outcomes of laparoscopic donor nephrectomy with multiple renal arteries. Int Braz J Urol. 2012 Jul-Aug;38(4):496-503. doi: 10.1590/s1677-55382012000400009. PMID 22951178
- [Background] Simforoosh N, Basiri A, Tabibi A, Shakhssalim N, Hosseini Moghaddam SM. Comparison of laparoscopic and open donor nephrectomy: a randomized controlled trial. BJU Int. 2005 Apr;95(6):851-5. doi: 10.1111/j.1464-410X.2005.05415.x. PMID 15794797
- [Background] Hoda MR, Hamza A, Greco F, Wagner S, Fischer K, Fornara P. Early and late graft function after laparoscopic hand-assisted donor nephrectomy for living kidney transplantation: comparison with open donor nephrectomy. Urol Int. 2010;84(1):61-6. doi: 10.1159/000273468. Epub 2010 Feb 17. PMID 20173371
- [Background] Fonouni H, Mehrabi A, Golriz M, Zeier M, Muller-Stich BP, Schemmer P, Werner J. Comparison of the laparoscopic versus open live donor nephrectomy: an overview of surgical complications and outcome. Langenbecks Arch Surg. 2014 Jun;399(5):543-51. doi: 10.1007/s00423-014-1196-4. Epub 2014 Apr 28. PMID 24770877
- [Background] Nanidis TG, Antcliffe D, Kokkinos C, Borysiewicz CA, Darzi AW, Tekkis PP, Papalois VE. Laparoscopic versus open live donor nephrectomy in renal transplantation: a meta-analysis. Ann Surg. 2008 Jan;247(1):58-70. doi: 10.1097/SLA.0b013e318153fd13. PMID 18156924
- [Background] Ungbhakorn P, Kongchareonsombat W, Leenanupan C, Kijvikai K, Wisetsingh W, Patcharatrakul S, Jirasiritam S. Comparative outcomes of open nephrectomy, hand-assisted laparoscopic nephrectomy, and full laparoscopic nephrectomy for living donors. Transplant Proc. 2012 Jan;44(1):22-5. doi: 10.1016/j.transproceed.2011.12.026. PMID 22310568
- [Background] Jacobsson A, Nedergaard J, Cannon B. alpha- and beta-adrenergic control of thermogenin mRNA expression in brown adipose tissue. Biosci Rep. 1986 Jul;6(7):621-31. doi: 10.1007/BF01114756. PMID 3022838
- [Background] Garcia-Garcia G, Renoirte-Lopez K, Marquez-Magana I. Disparities in renal care in Jalisco, Mexico. Semin Nephrol. 2010 Jan;30(1):3-7. doi: 10.1016/j.semnephrol.2009.10.001. PMID 20116641
- [Background] Mallafre Sala JM. [Living donor nephrectomy for kidney transplantation]. Arch Esp Urol. 2005 Jul-Aug;58(6):517-20. doi: 10.4321/s0004-06142005000600008. Spanish. PMID 16138763
- [Background] Fabian JF, Mancilla E, Aburto JS, Kasep J, Lopez JO, Almaguer F, Basilio CI, Garcia HB, Arcos AG. Hand-Assisted Laparoscopic Nephrectomy for Live Donor Kidney Transplantation. Transplant Proc. 2016 Mar;48(2):568-71. doi: 10.1016/j.transproceed.2016.02.020. PMID 27110004
- [Background] Greco F, Hoda MR, Alcaraz A, Bachmann A, Hakenberg OW, Fornara P. Laparoscopic living-donor nephrectomy: analysis of the existing literature. Eur Urol. 2010 Oct;58(4):498-509. doi: 10.1016/j.eururo.2010.04.003. Epub 2010 Apr 18. PMID 20417024
- [Background] Alfonzo JP. Four decades of kidney transplantation in Cuba. MEDICC Rev. 2013 Jan;15(1):23-8. doi: 10.37757/MR2013V15.N1.6. PMID 23396238
- [Background] Matevossian E, Kern H, Huser N, Doll D, Snopok Y, Nahrig J, Altomonte J, Sinicina I, Friess H, Thorban S. Surgeon Yurii Voronoy (1895-1961) - a pioneer in the history of clinical transplantation: in memoriam at the 75th anniversary of the first human kidney transplantation. Transpl Int. 2009 Dec;22(12):1132-9. doi: 10.1111/j.1432-2277.2009.00986.x. No abstract available. PMID 19874569
- [Background] Barker CF, Markmann JF. Historical overview of transplantation. Cold Spring Harb Perspect Med. 2013 Apr 1;3(4):a014977. doi: 10.1101/cshperspect.a014977. PMID 23545575
- [Background] Wilson CH, Sanni A, Rix DA, Soomro NA. Laparoscopic versus open nephrectomy for live kidney donors. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD006124. doi: 10.1002/14651858.CD006124.pub2. PMID 22071829
- [Background] Cabral JF, Braga I, Fraga A, Castro-Henriques A, Principe P, Silva-Ramos M. From Open to Laparoscopic Living-donor Nephrectomy: Changing the Paradigm in a High-volume Transplant Center. Transplant Proc. 2015 May;47(4):903-5. doi: 10.1016/j.transproceed.2015.03.037. PMID 26036482